CLINICAL TRIAL: NCT03268655
Title: Pilot Trial to Examine the Effect of Ginger on the Gut Microbiome (GINGER)
Brief Title: Ginger and Gut Microbiome (GINGER)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SPH-2017-25928; Anna-CPRC-TBD (Other: UMN Clinical Protocol Review Committee)
Record Dates: First submitted 2017-08-25; First posted 2017-08-31 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Adenoma
Keywords: gingerol; microbiome; gut; ginger
MeSH Terms: interventions — ginger extract

STUDY DESIGN:
Intervention Model Description: Pilot. Double-blind placebo-controlled randomized trial
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginger extract (Experimental): Ginger extract, 2000 mg daily for 6 weeks, followed by 6 week washout.
  Interventions: Dietary Supplement: Ginger extract
- Placebo (Experimental): Placebo, daily for 6 weeks, followed by 6 week washout.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ginger extract — 2000 mg ginger extract daily for 6 weeks, plus 6 weeks washout
  Arms: Ginger extract
Other: Placebo — 2000 mg ginger extract daily for 6 weeks, plus 6 weeks washout
  Arms: Placebo

SUMMARY:
Estimate the impact of a 6-week daily intake of 2000 mg of ginger extract on the composition of the gut microbiome using a randomized placebo-controlled double-blinded design, i.e. examine the change of microbiome over time within and between the subjects..

DETAILED DESCRIPTION:
This is a pilot trial to evaluate the feasibility of conducting a large randomized trial and estimate the effects of ginger extract on the gut microbiome. The pilot study will recruit from multiple sites 95-100 subjects aged 50-75 years old who were diagnosed with colorectal adenoma within the last five years. There will be 47-50 subjects in the treatment group and 47-50 in the placebo group. The subjects will be randomized to receive either 2000 mg of ginger extract per day (1000 mg twice a day) or matching placebo.

Subjects will provide three stool specimens for analysis of the intestinal microbiome over a 12-week period at the following intervals: Week 0 (Day 1), Week 6, and Week 12. Although the gut microbiome is stable within a period of 1-2 months, a control arm will be included to account for potential dietary and other changes that may affect the gut microbiome. Gut microbiome composition - the presence, abundance, and diversity of bacterial taxa - will be derived by sequencing microbial 16S ribosomal RNA genes.

Primary Aims:

Aim 1 is to estimate the impact of a 6-week daily intake of 2000 mg of ginger extract on the composition of the gut microbiome using a randomized placebo-controlled double-blinded design, i.e. examine the change of microbiome over time within and between the subjects.

Aim 2 will examine the correlation between the ginger-related changes in microbiome profile with the levels of circulating biomarkers: urinary Prostaglandin E (PGE) metabolites.

Hypothesis: In the ginger versus placebo arm, gut microbiome will shift towards a lower proportion of pro-inflammatory, bacteria associated with colorectal cancer (CRC) and higher proportion of anti-inflammatory, CRC-protective bacteria.

Secondary Aim:

1. At the end of the study, we expect to show that ginger decreases the relative abundance of pro-inflammatory, CRC-predisposing taxa and increases the abundance of anti-inflammatory, CRC-protective taxa, i.e., demonstrate that ginger boosts changes in gut microbiome that are protective against CRC, as well as assess ginger-induced changes in immune response.
2. The similarities of bacterial profiles will be compared between three time points baseline and 6 Weeks and 12 Weeks to estimate whether 6-week is a sufficient time for washout.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal adenoma diagnosis

Exclusion Criteria:

* Allergy or sensitivity to ginger
* Active cancer
* Unstable medical condition
* Unstable diet or weight

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Composition of the gut microbiome | Baseline to 6 Weeks
  Fecal microbial diversity and the prevalence of specific taxa associated with colorectal cancer (e.g. Fusobacteria, butyrate producing bacteria) will be estimated at 6 weeks. The ginger-related changes in the prevalence of each taxon will be assessed individually and also combined into a microbiome index (the abundance of protective taxa will be included as a negative value).
Urine inflammatory biomarker | Baseline to 6 weeks
  Urinary metabolite of Prostaglandin E2 (ng/mg of creatinine) will be measured before and after treatment with ginger. Changes in inflammatory markers will be correlated to changes in the microbial diversity and the microbiome composition

SECONDARY OUTCOMES:
Change in gut microbiome composition | Baseline to 12 weeks
  Beta-diversity will be compared between three time points: baseline, 6 Weeks and 12 Weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Prizment, PhD, MPH, Principal Investigator — University of Minnesota, Epidemiology and Community Health
Locations (13):
- United States (13):
  - Mayo Clinic Cancer Center, Albert Lea, Minnesota
  - Mayo Clinic Cancer Center, Austin, Minnesota
  - Essentia Health - Deer River, Deer River, Minnesota
  - Essentia Health St Mary's - Detroit Lakes, Detroit Lakes, Minnesota
  - Essentia Health - Fosston Clinic, Fosston, Minnesota
  - Fairview Grand Itasca Clinic & Hospital, Grand Rapids, Minnesota
  - Fairview Range Medical Center, Hibbing, Minnesota
  - Mayo Clinic Cancer System, Mankato, Minnesota
  - Epidemiology Clinical Research Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Park Rapids Clinic, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - Essentia Health -Virgina Clinic, Virginia, Minnesota

IPD SHARING:
Plan to Share IPD: No
The results of the study will be disseminated to various stakeholders through the publication of a manuscript in a peer-reviewed journal and through presentation at scientific meetings.